CLINICAL TRIAL: NCT02316028
Title: A Phase I Clinical Trial on Decitabine (5-aza-2'-Deoxycytidine) Administered by Hepatic Arterial Infusion in Patients With Unresectable Liver-predominant Metastases From Colorectal Cancer
Brief Title: Phase I:Decitabine by Hepatic Arterial Infusion(HAI) in Unresectable Liver Metastases Colorectal Cancer (CRC)
Acronym: DECIT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UZB-BN-2013-002
Record Dates: First submitted 2014-12-03; First posted 2014-12-12 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Liver Metastasis; Colorectal Cancer
Keywords: decitabine; colorectal cancer; hepatic arterial infusion
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- decitabine (Experimental): administration of decitabine by hepatic arterial infusion
  * Accrual of patients and dosing of decitabine will be guided by a traditional 3+3 design using an accelerated titration for the first three dose levels.
  * Proposed dose levels:
    1. 10 mg/m2 per course
    2. 15 mg/m2 per course
    3. 20 mg/m2 per course
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — administration of decitabine by hepatic arterial infusion
  * Accrual of patients and dosing of decitabine will be guided by a traditional 3+3 design using an accelerated titration for the first three dose levels.
  * Proposed dose levels:
    1. 10 mg/m2 per course
    2. 15 mg/m2 per course
    3. 20 mg/m2 per course
  Other Names: Dacogen

SUMMARY:
Despite the advances in the medical treatment of unresectable liver metastases from colorectal cancer there is currently no curative treatment option available for these patients. Decitabine is a cytidine analog with proven anti-neoplastic activity in patients with acute myeloid leukemia and myelodysplastic syndromes. Decitabine causes demethylation of the DNA strands of replicating cells. Hereby decitabine treatment demethylates the promoter regions of tumor suppressor- and cancer testis antigen encoding genes leading to expression of these genes by the cancer cells. The hepatic arterial route for administration of cytotoxic drugs has been widely explored in treatment of colorectal cancer liver metastases because these metastases depend for their blood flow from this artery (as opposed to the normal liver tissue that is mainly dependent from the portal vein). By investigating the administration of decitabine by hepatic arterial infusion the investigators intend to explore the potential advantage of minimizing the systemic exposure (and toxicity) and maximizing the concentration of decitabine within the liver metastasis. The primary objective of this phase I will be to establish the recommended dose for decitabine by HAI for further use in phase II trials. The most important secondary objective will be to document the effect of decitabine by HAI on the expression of cancer testis antigens by the colorectal cancer cells, serving as a reference for potential further exploration of decitabine by HAI in combination with cancer immunotherapy

DETAILED DESCRIPTION:
This clinical trial will recruit eligible patients diagnosed with unresectable liver-predominant colorectal cancer metastases who have experience progression of their disease following standard of care treatment.

Unless patients already dispose of a hepatic arterial catheter, they will undergo placement of a permanent hepatic artery catheter (by laparoscopic surgery). During this surgical procedure a biopsy will be made of the colorectal cancer liver metastasis.

Decitabine will be administered as a daily 1-hour IV infusion on 5 consecutive days, every 4weeks.

Two weeks after the first day of administration of decitabine, a CT-guided biopsy a liver metastasis will be performed in order to obtain tumor tissue for histopathological analysis and DNA/RNA extraction for the purposes of methylation specific Polymerase Chain Reaction (PCR) and reverse transcriptase PCR for assessment of demethylation and expression of cancer-testis antigen encoding genes.

Blood samples for collection of "cell-free DNA" and White Blood Cell (WBC ) for the purpose of DNA/RNA extraction and analysis by methylation specific PCR and reverse transcriptase PCR for assessment of demethylation and expression of cancer-testis antigen encoding genes will be obtained weekly after decitabine treatment.

The dose of decitabine will be escalated in subsequent patient cohorts enrolled to this phase I trial (see rules for dose escalation).

Study treatment will be continued until unacceptable toxicity, progressive disease or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of colorectal adenocarcinoma CRC stage IV with predominant unresectable liver metastases and at least one measurable metastatic liver lesion
* Performance status WHO criteria of < 2.
* Laboratory values: absolute neutrophil count (ANC) count > 1500 /mm³, Platelet count > 100 000 /mm³, Lymphocytes > 800 /mm³, Serum creatinine < 2.0 mg/dl or creatinine clearance >40 ml/min, Serum bilirubin < 2.0 mg/dl
* Progressive disease following standard of care palliative systemic chemotherapy
* able to give written informed consent.

Exclusion Criteria:

* No prior radiotherapy to all target liver lesions
* No previous history of gastric or hepatobiliary surgery (except for simple cholecystectomy, No concurrent liver disease or other serious medical disease or condition
* No concomitant use of other investigational drugs.
* No pre-existing neuropathy with a severity of > grade 1 in the WHO toxicity scale.
* No previous or concurrent malignancies except for adequately treated in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma of the skin or any other malignancy given potentially curative treatment more than 5 years before study entry
* No pregnant or breast-feeding female patients, use of an effective contraceptive if the risk of conception exists during study treatment.
* No candidate for the resection of all CRC metastases with curative intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
toxicity of escalating doses of decitabine administered by HAI | 2years
  : to establish the recommended dose of decitabine administered by hepatic arterial infusion in patients with unresectable liver-predominant metastases from colorectal cancer

SECONDARY OUTCOMES:
overall survival | 5years
  overall survival
progression free survival | 5 years
  progression free survival
best objective tumor response | 5 years
  Best objective tumor response (BOR) per Response Evaluation Criteria in Solid Tumors (RECIST ), version 1.1
measuring Global DNA methylation of tumoral DNA | 2years
  Determine the methylation status of the promoter region and messenger ribonucleic acid (mRNA) expression of cancer-testis antigens in pré- and post treatment biopsies of colorectal cancer liver metastases
measuring Global DNA methylation of cell free DNA | 2years
  Determine the ratio of demethylated versus methylated DNA corresponding to the promoter region of cancer-testis antigen encoding genes on the circulating free DNA (cfDNA) in venous blood prior to and following the administration of decitabine by HAI

CONTACTS AND LOCATIONS:
Overall Officials: Bart Neyns, PhD, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - UZ Brussel, Jette, Brabant
  - UZ Brussel, Brussels

REFERENCES:
- [Derived] Jansen YJL, Verset G, Schats K, Van Dam PJ, Seremet T, Kockx M, Van Laethem JB, Neyns B. Phase I clinical trial of decitabine (5-aza-2'-deoxycytidine) administered by hepatic arterial infusion in patients with unresectable liver-predominant metastases. ESMO Open. 2019 Mar 5;4(2):e000464. doi: 10.1136/esmoopen-2018-000464. eCollection 2019. PMID 30962963